CLINICAL TRIAL: NCT06020508
Title: Pilot Study for Human Clinical Trial to Evaluate the BRIGHTPOINT Reflectometer Device as Secondary Confirmation to Loss of Resistance in Lumbar Epidural Placement
Brief Title: Lumoptik BRIGHTPOINT Reflectometer Device for Lumbar Epidural Placement
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0074
Record Dates: First submitted 2023-08-28; First posted 2023-08-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Lumbar Spine Surgery
Keywords: epidural; neuraxial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Group 1: Attending anesthesiologists who are trained in epidural placement will perform neuraxial procedures (CSEs, Epidural, Spinals through an epidural needle) utilizing loss of resistance with saline in conjunction with the Lumoptik BrightPoint Epidural Device. The Lumoptik device will be connected between a standard commercially available 17G or 18G, 3.5-inch epidural needle and a saline filled loss of resistance syringe. The anesthesiologist will view the Lumoptik BrightPoint visual display in real time as the epidural procedures are performed. The LOR epidural procedure using haptic feedback will be used as the primary confirmation of correct needle placement in the epidural space. Graphic and color circle information from the Lumoptik visual display will be used as a secondary confirmation of epidural placement.
  Interventions: Device: Group 1 - Lumoptik BrightPoint Epidural Device

INTERVENTIONS:
Device: Group 1 - Lumoptik BrightPoint Epidural Device — Participants will undergo a neuraxial procedure to measure loss of resistance with saline in conjunction with the Lumoptik BrightPoint Epidural Device.

SUMMARY:
The goal of this clinical trial is to test the BrightPoint Epidural device as the first system to use multispectral reflectometry to find the epidural space in lumbar neuraxial procedures requiring epidural needle. The main questions it aims to answer are:

1. Is the device a qualitatively effective secondary confirmation of Loss of Resistance?
2. Is the device a qualitatively effective training tool for educating trainees in how to perform lumbar epidurals?

Participants will undergo a neuraxial procedure in which the attending anesthesiologist will use the BrightPoint epidural device to form an opinion on its effectiveness in confirming epidural space access.

DETAILED DESCRIPTION:
There have been few improvements to the LOR technique from a device standpoint in recent years, and those that options do exist have not achieved widespread clinical use. The devices that do exist are variations on pressure sensors, some automate the "resistance" by placing various systems in place to apply a pressure to the plunger so that it will inject when the epidural space is accessed without the practitioner doing it themselves. This concept is represented by devices such as the Epimatic syringe from Vygon. Others improve on this concept by monitoring the pressure required to inject a set volume of fluid, thus being able to differentiate between true and false losses, as during false losses the pressure will increase as more fluid is injected. This system is represented by the CompuFlo Device by Milestone Scientific.

The BrightPoint Epidural device is the first system that utilizes multispectral reflectometry in order to identify the epidural space. This technology has the theoretical benefit over pressure-based systems of being able to identify and differentiate between different issue types (muscle, ligament, bone) as the needle is advanced towards the epidural space. Lumoptik, the company behind the BrightPoint Epidural device, is an early-stage startup based in Cleveland, Ohio. The main questions this trial aims to answer are:

1. Is the device a qualitatively effective secondary confirmation of Loss of Resistance?
2. Is the device a qualitatively effective training tool for educating trainees in how to perform lumbar epidurals?

This trial is being conducted to improve our current standard of care in neuraxial placement of loss-of-resistance. While the loss of resistance technique is tried and true, especially in experienced hands, complications such as dural punctures, misplaced epidurals, patchy epidurals, neurologic injuries, and intravascular catheters can occur even in experienced hands. All of which can cause significant patient morbidity and costs to the healthcare system, and as is shown in the Lacombe attached, the effects of dural puncture can be long lived for the patient. There can also be a steep learning curve when learning the technique, with the frequency of inadvertent dural punctures significantly higher in the early stages of learning the procedure. Therefore, we as a specialty are obligated to evaluate potential improvements to our current way of practice to reduce the burden to our patients from the complications of our interventions.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing a lumbar neuraxial procedure requiring epidural needle
* Age 18-99

Exclusion Criteria:

* Previous lumbar spine surgery
* Any known spinal abnormality that would interfere with successfully advancing a needle into the epidural space
* Any patient requiring epidural needle longer than 4 inches
* Any contraindication to neuraxial anesthesia
* Tattoo at the site of epidural insertion

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to have surgery at the Hospital for Special Surgery that will require a lumbar neuraxial procedure requiring an epidural needle.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Real time confirmation of epidural space with loss of resistance technique | Post-operation (after the surgery is complete)
  On the post-procedure questionnaire, the anesthesiologist will report about whether the device identified epidural space in agreement with loss of resistance technique.
  If no, the outcome will be recorded as either a false positive (device signaled epidural space while needle was not in epidural space) or false negative (device did not signal epidural space while needle was in epidural space).

SECONDARY OUTCOMES:
Clinical (anesthesiologist) opinions on Lumoptik Bright Point Epidural device | Post-operation (after the surgery is complete)
  On the post-procedure questionnaire, the anesthesiologist will give their opinion about the device following their use of the study device.
Color graphics aid in the identification of needle tips. | Post-operation (after the surgery is complete)
  On the post-procedure questionnaire, the proceduralist will give a yes or no answer to the prompt to the question "Did the Bright Point Epidural color graphic improve your understanding of where your needle tip is or what tissue it is in?"
The time it takes to insert the epidural needle into the patient's skin. | From "in OR time" to "time when needle is inserted"
  The time between when the patient entered the operating room and when the epidural needle was inserted into the patient's skin.
The time it takes to successfully identify the epidural space. | From "time when needle is inserted" to "time when epidural space is identified"
  The time between inserting an epidural needle into the skin and successfully identifying the epidural space.
The percentage of Successful Neuraxial Procedures | Post-operation (after the surgery is complete)
  The percentage of successful neuraxial procedures, calculated by dividing "the number successful neuraxial procedures placed without assistance or complication by the number of attempted neuraxial procedures"

CONTACTS AND LOCATIONS:
Overall Officials: Michael Singleton, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lacombe A, Downey K, Ye XY, Carvalho JCA. Long-term complications of unintentional dural puncture during labor epidural analgesia: a case-control study. Reg Anesth Pain Med. 2022 Jun;47(6):364-369. doi: 10.1136/rapm-2021-103266. Epub 2022 Mar 25. PMID 35338103
- [Result] van der Hek H, Plomp HN. Occupational stress management programmes: a practical overview of published effect studies. Occup Med (Lond). 1997 Apr;47(3):133-41. doi: 10.1093/occmed/47.3.133. PMID 9156467